CLINICAL TRIAL: NCT01311596
Title: Show Me to Help Me
Status: Completed | Type: Observational
Sponsor: Akron Children's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 101201
Record Dates: First submitted 2011-03-08; First posted 2011-03-09 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Autism
Keywords: icons in clinic or office for patients with Autism
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- No icons: Clinic - Children who are established patients, 4-18 years old, and presented to the NeuroDevelopmental Science Center for a follow-up office visit during the first 2 weeks of the study period
  Lab -Patients 4-18 years old with a documented diagnosis who were seen in the NeuroDevelopmental Science Center and were given a prescription for lab work during the first 2 weeks of the study period
- Icons: Clinic - Children who are established patients, 4-18 years old, and presented to the NeuroDevelopmental Science Center for a follow-up office visit during the last 2 weeks of the study period
  Lab - Patients 4-18 years old with a documented diagnosis who were seen in the NeuroDevelopmental Science Center and were given a prescription for lab work during the last 2 weeks of the study period
  Interventions: Other: Icons

INTERVENTIONS:
Other: Icons — Clinic- patients first shown picture icons of the steps of taking vital signs Lab - patients first shown picture icons of the steps of a blood draw procedure
  Other Names: Picture Exchange communication system (PECS)
  Groups: Icons

SUMMARY:
This cohort observation, randomized controlled trial is intended to provide data that icons and non-verbal communication improve communication and cooperation with children with Autism/communication delay and aid in the transition to an unfamiliar environment. It would lay the foundation for future studies and practices of using icons and pictures for the whole office visit to enhance communication between the patient and physician/nurse/medical staff and cooperation of the patient.

1. Use icons during triage/check in process to decrease time and increase patient compliance. Compare typical children to those with Autism/communication delay.
2. Use icons during blood draw to improve communication with patients, to help with patient understanding, and increase patient cooperation and decrease noise and length of procedure.

ELIGIBILITY:
Inclusion Criteria:

* established patients with a documented diagnosis
* 4-18 years old
* present to the NeuroDevelopmental Center during the study period
* Lab study: given prescription for lab work that will be following the visit or the next day in the Locust outpatient lab

Exclusion Criteria:

* <4 years old or >18 years old
* new patient
* diagnosis not documented
* Lab study: lab work will be drawn at another lab or more than 1 day later

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children who are established patients, 4-18 years old, and present to the NeuroDevelopmental Science Center for a follow-up office visit during the study period, since a diagnosis will be available at the time of the study (patients in the lab study may be new patients if they have a diagnosis at the time their lab work is prescribed). The NeuroDevelopmental Science Center at Akron Children's Hospital provides nearly 25,000 visits annually to children and youth affected by neurological, developmental, and behavioral disorders. This includes children with autism, intellectual disabilities, physical disabilities, learning disabilities, epilepsy and other neurological conditions.
Sampling Method: Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2011-02; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Icons improve understanding, transition and cooperation of the child with Autism/communication delay as measured by improved times for the obtainment of vital signs | 4 weeks

SECONDARY OUTCOMES:
Icons improve understanding and cooperation of the child with Autism/communication delay as measured by improved times of lab draws, success of lab draws, and decreased noise level | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Akron Children's Hospital, Akron, Ohio, United States

REFERENCES:
- [Background] Bondy A, Frost L. The Picture Exchange Communication System. Behav Modif. 2001 Oct;25(5):725-44. doi: 10.1177/0145445501255004. PMID 11573337
- [Background] Charlop-Christy MH, Carpenter M, Le L, LeBlanc LA, Kellet K. Using the picture exchange communication system (PECS) with children with autism: assessment of PECS acquisition, speech, social-communicative behavior, and problem behavior. J Appl Behav Anal. 2002 Fall;35(3):213-31. doi: 10.1901/jaba.2002.35-213. PMID 12365736
- [Background] Desch LW, Gaebler-Spira D; Council on Children With Disabilities. Prescribing assistive-technology systems: focus on children with impaired communication. Pediatrics. 2008 Jun;121(6):1271-80. doi: 10.1542/peds.2008-0695. PMID 18519500
- [Background] Francis K. Autism interventions: a critical update. Dev Med Child Neurol. 2005 Jul;47(7):493-9. doi: 10.1017/s0012162205000952. PMID 15991872
- [Background] Ganz JB, Simpson RL. Effects on communicative requesting and speech development of the Picture Exchange Communication System in children with characteristics of autism. J Autism Dev Disord. 2004 Aug;34(4):395-409. doi: 10.1023/b:jadd.0000037416.59095.d7. PMID 15449515
- [Background] Magiati I, Howlin P. A pilot evaluation study of the Picture Exchange Communication System (PECS) for children with autistic spectrum disorders. Autism. 2003 Sep;7(3):297-320. doi: 10.1177/1362361303007003006. PMID 14516062
- [Background] Sulzer-Azaroff B, Hoffman AO, et al. The Picture Exchange Communication System (PECS): What Do the Data Say? Focus on Autism and Other Developmental Disabilities. 209;24(2):89-103